CLINICAL TRIAL: NCT01706835
Title: An Open-Lable Phase 1 Study to Investigate the Pharmacolkinetics of Aldoxorubicin (INNO-206;DOXO-EMCH) Administered as a 30 Minute Infusion Every 3 Weeks in Subjects With Advanced Solid Tumors
Brief Title: Study to Investigate the Pharmacolkinetics of Aldoxorubicin (INNO-206;DOXO-EMCH) Administered as a 30 Minute Infusion Every 3 Weeks in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P1-PK-01
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2014-12

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumor; aldoxorubicin; phase 1; pharmacokinetic; INNO-206
MeSH Terms: interventions — DOXO-EMCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aldoxorubicin (Experimental): Aldoxorubicin dosages of 230 mg/m2 or 350 mg/m2 will be given as a 30 minute infusion every 3 weeks for 8 cycles.
  Interventions: Drug: aldoxorubicin

INTERVENTIONS:
Drug: aldoxorubicin
  Other Names: INNO-206

SUMMARY:
This is a phase 1 open-label study to investigate the pharmacokinetics of aldoxorubicin administered as a 30 minute infustion every 3 weeks for up to 8 cycles in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
An Open-Label Phase 1 Study to Investigate the Pharmacokinetics of Aldoxorubicin Administered as a 30 Minute Infusion Every 3 Weeks in Subjects with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Histologically or cytologically confirmed malignant solid tumor that has relapsed or is refractory to standard therapy.
3. Subjects who have received prior radiation therapy with stable central nervous system (CNS) metastasis with no progression of brain metastasis by CT/MRI scan in last 4 weeks.
4. Capable of providing informed consent and complying with trial procedures.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2.
6. Life expectancy >12 weeks.
7. Measurable or evaluable disease.
8. Women must not be able to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. [Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.].
9. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
10. Geographic accessibility to the site.

Exclusion Criteria:

1. Palliative surgery, chemotherapy, immunotherapy and/or radiation treatment less than 4 weeks prior to the Screening Visit.
2. Exposure to any investigational agent within 30 days of the Screening Visit.
3. Laboratory values: Screening serum creatinine greater than or equal to 1.5 mg/dL, alanine aminotransferase (ALT) greater than 3 times the upper limit of normal (ULN) or 5 times the ULN in liver metastases, total bilirubin greater than 3 times the ULN, white blood cell (WBC) count <3500/mm3, absolute neutrophil (ANC) count < 2000/mm3, platelet concentration <100,000/mm3, hematocrit level <25% for females or <28% for males (transfusion is allowed during screening).
4. Clinically evident congestive heart failure (CHF) > class II of the New York Heart Association (NYHA) guidelines.
5. Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
6. Recent history (within 6 months) or current signs of active coronary artery disease with or without angina pectoris.
7. Serious myocardial dysfunction defined scintigraphically (MUGA, myocardial scintigram) or ultrasound determined absolute left ventricular ejection fraction (LVEF) <45% of predicted.
8. Known history of HIV infection.
9. Active, clinically significant serious infection requiring treatment with antibiotics, antivirals or antifungals.
10. Major surgery within 4 weeks prior to treatment.
11. Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
12. Any condition that is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | up to 3 months
  Blood samples will be obtained for pharmacokinetics. Standard pharmacokinetic parameters, including t1/2, Cmax, AUC, Vd and CL, will be determined.

SECONDARY OUTCOMES:
Safety | up to 6 months
  All subjects who receive any amount of aldoxorubicin will be included in the safety analyses, which will include the following:
  1. The incidence, severity, duration, causality, seriousness, and type of AEs and changes in the subject's physical examination, vital signs, and clinical laboratory results.
  2. Deaths and other SAEs will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levitt, MD, Study Director — CytRx Coorporation
Locations (1):
- Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California, United States